CLINICAL TRIAL: NCT01469247
Title: Phase I/II Study of Reirradiation of Recurrent or Progressive Brainstem Glioma
Brief Title: Diffuse Intrinsic Pontine Glioma (DIPG) Reirradiation (ReRT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0804; NCI-2011-03725 (Registry Identifier: NCI CTRP); R01CA187202 (NIH)
Record Dates: First submitted 2011-11-04; First posted 2011-11-10 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Brain Cancer
Keywords: Brain cancer; Recurrent or progressive brainstem glioma; Diffuse Intrinsic Pontine Glioma; DIPG; Reirradiation; ReRT; Photon radiation therapy; XRT
MeSH Terms: conditions — Brain Neoplasms; Recurrence; Diffuse Intrinsic Pontine Glioma | interventions — Radiotherapy; Re-Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation Therapy (Experimental): Starting dose of 24 Gray (Gy) in 2 Gy fractions.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Starting Dose 24 Gy in 2 Gy fractions.
  Other Names: XRT; Reirradiation

SUMMARY:
The goal of this clinical research study is to find a safe dose of radiation that can be given to patients with brainstem glioma who have already received radiation therapy.

You will receive photon radiation therapy. This type of radiation is similar to the radiation you have already had. Conformal radiotherapy or intensity modulated radiotherapy (IMRT) will be used to try to treat the tumor while affecting as little of the surrounding normal tissue as possible.

DETAILED DESCRIPTION:
Radiation Therapy Administration:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of radiation therapy based on when you join this study. Three (3) dose levels of radiation therapy will be tested. Three (3) participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will be randomly assigned (as in the roll of dice) to one of the dose levels, and the assignment will also depend on how the previous participants have done. Participants will not be assigned to one of the higher 2 of the 3 dose levels unless the lower dose level is found to be tolerable. The first and second groups will receive 12 treatments and the third group will receive 14 treatments (Monday through Friday for about 2½ weeks). Your doctor will tell you how many treatments you will receive.

You may be given drugs to help prevent side effects. The study staff will tell you about these drugs, how they will be given, and the possible risks.

Study Visits:

About 2-4 days before you start radiation therapy, you will have a simulation. During the simulation session, a mask will be made of your face and head to keep you still. You will also have a computed tomography (CT) scan. This process allows the radiation planning to take place. Sedation by an anesthesiologist (anesthesia doctor) will be used if needed for young children to allow the radiotherapy to be delivered safely.

One (1) time a week for 3 weeks, and then 1 time a month (30 days +/- 10 days) for 2 months or unless the disease gets worse:

* You will have a neurological exam.
* Your performance status will be recorded.
* You will fill out the quality-of-life questionnaire.
* You will be asked about any side effects you may have had.

You will have a magnetic resonance imaging (MRI) scan of the brain within 1 month after joining the study.

Length of Treatment:

You may continue receiving radiation therapy for 12 or 14 treatments. You will no longer be able to receive radiation therapy if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Follow-up Visits:

One (1) month after you finish radiation therapy, at 6-8 weeks, then every 2-3 months after that from then on, you will have an MRI scan to check the status of the disease. The MRI scan will include advanced imaging to learn if the tumor has come back or if there is brain tissue damage from the radiation. With this type of imaging, a temporary infusion line with a bigger than standard size needle will be inserted to your vein if you do not already have a power port-a-cath in place. This may take between 20-30 minutes.

This is an investigational study. Radiation therapy in this study is delivered using FDA-approved and commercially available methods. It is investigational to find the best dose of radiation therapy to use for repeat radiation therapy.

Up to 30 participants will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of DIPG by MRI imaging defined as tumor that has a pontine epicenter and is diffuse (tumor that involves the majority (>50%) of the brainstem) on T2 or FLAIR imaging rather than focal. Histologic confirmation is not required
2. Radiation therapy to brain for DIPG that was completed at least 10 months prior to planned reirradiation
3. Clinical progression of symptoms with any radiographic progression on MRI within 21 days prior to registration (any progression in size or enhancement on MRI along with worsening symptoms, will be defined as progression prior to enrollment). Radiographic progression is defined as any increase in tumor size (in axial or sagittal images) or progressive contrast enhancement and abnormal T2/FLAIR signal by MRI.
4. Signed informed consent by patient and/or parents or legal guardian
5. Lansky/Karnofsky Performance Status score of 40-100
6. Central nervous system function defined as not severely somnolent or comatose (central cortical neurotoxicity scale <Grade 3)
7. Life expectancy of >/= 8 weeks

Exclusion Criteria:

1. Prior radiation of greater than 60 Gy to >20% of brainstem.
2. Patients with Neurofibromatosis 1 because the biologic behavior of their tumors may be more benign
3. Asymptomatic patients because the primary goal of treatment is palliation of symptoms
4. Pregnancy

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2011-12-07 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Optimal Dose Level Among Three Radiation Therapy (RT) Dose Levels | 1 month after radiation therapy
  Optimal dose level among three RT dose levels, defined in terms of the biologically equivalent dose (BED). The BED is given by the formula BED = (Total Dose)*(1 + d/3), denoting d = dose/fraction, with the constant 3 corresponding to brain tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Susan L. McGovern, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Orlando Health, Orlando, Florida
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org